CLINICAL TRIAL: NCT00859170
Title: Use of the Accordion Stone Management Device in Laser Lithotripsy
Brief Title: Use of Antiretropulsion Device in Laser Lithotripsy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in priorities occurred
Sponsor: Percutaneous Systems, Inc. (Industry)
Responsible Party: Thomas Lawson, PhD / VP, Clinical & Regulatory Affairs, Percutaneous Systems, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 08-001
Record Dates: First submitted 2009-03-05; First posted 2009-03-10 (Estimated); Last update posted 2010-01-08 (Estimated); Status verified 2010-01

CONDITIONS: Kidney Stones
Keywords: kidney stones; ureter; laser lithotripsy
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Accordion use (Experimental): Use of an Accordion device during the lithotripsy.
  Interventions: Device: Accordion device
- Control Group (No Intervention): Patients who will not have an Accordion device used during lithotripsy.

INTERVENTIONS:
Device: Accordion device — an antiretropulsion device
  Other Names: Accordion Stone Management Device PA1205-06-10
  Arms: Accordion use

SUMMARY:
The objectives of this post-market evaluation are

1. to assess the capacity of the procedure to be completed with use of only a semi-rigid ureteroscope, without requiring use of a flexible ureteroscope
2. to compare the rate of retropulsion and the time required to complete the lithotripsy in patients in which the Accordion device is used in contrast to when such a device is not employed.

DETAILED DESCRIPTION:
In North America, ureteroscopic-guided lithotripsy with the holmium:yttrium-aluminum-garnet (Ho:YAG) laser has increased in clinical utility owing to its capacity to fragment stones of all compositions. However, with the application of the light energy, retropulsion of the stone is possible due to the combined effects of fragment ejection, water vaporization, and cavitation bubble expansion then collapse. Reducing the laser energy and using laser fibers with small diameters are options to address such a consequence, but these changes have the potential to reduce the efficacy of the laser treatment.

Movement of stones and stone fragments during laser lithotripsy also can be caused by the application of irrigation during the procedure. Irrigation is necessary in order to maintain clear visualization of the targeted stone during lithotripsy, and yet irrigation flow pressure can push stones away from the laser tip, requiring repositioning of the laser, and, in the presence of hydrodilation of the ureter, cause the stone to float up to the renal pelvis or into the kidney itself. In such a situation the physician may be required to use more specialized instruments, adding to the complexity and cost of the procedure. As a result, physicians monitor irrigation closely and will reduce the flow if retropulsion of the stone or fragments occurs.

Retropulsion of stones and stone fragments during laser lithotripsy has been reported in up to 24% of patients and can cause prolonged operative times due to near-constant repositioning of the laser fiber between firings, and as well as result in additional treatment methods, making available a flexible ureteroscope, with its associated costs, and additional cost associated with an extended procedure.

A novel occluding guidewire, the Accordion Stone Management Device, has been developed that can be advanced up the ureter and past the stone. Once past the stone, an occlusion film is engaged within the lumen of the ureter in order to limit retropulsion of the stone and its fragments, irrespective of the laser energy, flow rate of irrigation, or dilation of the ureter. Reduction of stone fragment movement has the potential to reduce operative time and increase stone-free rates within this population.

ELIGIBILITY:
Inclusion Criteria:

* Solitary ureteral stone in the distal or medial ureter, 10 mm in diameter or less, as demonstrated by preoperative CT or IVP imaging and are 18 years of age or older.

Exclusion Criteria:

* Patients will be excluded from this study if they have active urinary tract infection, or, if female, pregnant, or has clinical evidence of sepsis, or a single or nonfunctioning kidney, or coagulopathy, or congenital ureteral abnormality, or previous ureteral reimplantation, or presence of any degree of ureteral stricture distal to the stone, as determined before or during the procedure, or inability to sign informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-06 (Estimated); Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of retropulsion or migration of the stone or fragments | Two months

SECONDARY OUTCOMES:
Elapsed times for placing the safety guidewire | Two months
Fragmenting the stone into pieces no larger than 1 mm in size | Two months
Removing the fragments from the ureter | Two months
Procedure time | Two months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas T Lawson, PhD, Study Director — Percutaneous Systems, Inc.
Locations (3):
- United States (3):
  - Kaiser Permanente Bellflower Hospital, Downey, California
  - New York University Medical Center, New York, New York
  - USMD Hospital, Arlington, Texas

REFERENCES:
- [Result] Manohar T, Ganpule A, Desai M. Comparative evaluation of Swiss LithoClast 2 and holmium:YAG laser lithotripsy for impacted upper-ureteral stones. J Endourol. 2008 Mar;22(3):443-6. doi: 10.1089/end.2007.0288. PMID 18355139
- [Result] Bapat SS, Pai KV, Purnapatre SS, Yadav PB, Padye AS. Comparison of holmium laser and pneumatic lithotripsy in managing upper-ureteral stones. J Endourol. 2007 Dec;21(12):1425-7. doi: 10.1089/end.2006.0350. PMID 18186678
- [Result] Ilker Y, Ozgur A, Yazici C. Treatment of ureteral stones using Holmium:YAG laser. Int Urol Nephrol. 2005;37(1):31-4. doi: 10.1007/s11255-004-6084-3. PMID 16132755
- [Result] Maislos SD, Volpe M, Albert PS, Raboy A. Efficacy of the Stone Cone for treatment of proximal ureteral stones. J Endourol. 2004 Nov;18(9):862-4. doi: 10.1089/end.2004.18.862. PMID 15659920